CLINICAL TRIAL: NCT06969443
Title: Evaluation of Rehabilitation Practices in Patients Undergoing Invasive Mechanical Ventilation in French-speaking Critical Care Units
Brief Title: Evaluation of Rehabilitation Practices in the Intensive Care Unit
Acronym: REHALITE
Status: Recruiting | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: SRLF-012025; 2025-A00025-44 (Other: IDRCB)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Invasive Mechanical Ventilation; Rehabilitation Exercise of ICU Patients
Keywords: ICU; Rehabilitation; Mechanical ventilation; Observationnal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Rehabilitation Procedure — Rehabilitation procedure list :
  1. Passive limb mobilization
  2. Active (or active-assisted) limb mobilization
  3. Passive transfer to chair
  4. Active transfer to chair
  5. Sitting on edge of bed
  6. Standing table (or similar)
  7. Standing on legs
  8. Walking
  9. Cyclo-ergometer (bed or chair)
  10. Electrostimulation

SUMMARY:
This observational study aims to describe the number of rehabilitation procedures performed per patient during their stay in French-speaking adult intensive care units undergoing invasive mechanical ventilation (average rehabilitation ratio). The study aims to determine the actual rehabilitation ratio, i.e. the number of rehabilitation procedures divided by the number of critical care hospital days (censored at day 28 from the start of invasive mechanical ventilation), provided to patients undergoing invasive mechanical ventilation. The rehabilitation procedure will remain the same, and ICU teams will only record the number of procedures performed per day.

ELIGIBILITY:
Inclusion criteria:

* Foreseeable invasive ventilation lasting more than 48 hours.
* Included within the first five days of an intensive care stay.

Exclusion criteria:

* Participation in an interventional study on early rehabilitation in the ICU
* Moribund patient
* Pregnant or breastfeeding woman
* A person deprived of liberty by court order
* Not being affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mechanical ventilation (MV) via an endotracheal tube for less than five days, in French-speaking intensive care units in three countries (France, Belgium and Switzerland), in whom MV is scheduled to last more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation Ratio | On Day 28 of study participation
  Number of rehabilitation procedures per day divided by the number of ICU days (censored at D28 from the start of invasive mechanical ventilation)

CONTACTS AND LOCATIONS:
Locations (1):
- SRLF, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided